CLINICAL TRIAL: NCT05001581
Title: Massive and Irreparable Rotator Cuff Tears Treated by Arthroscopic Partial Repair and Partial Repair With Long Head of the Biceps Tendon Augmentation. Comparison of Clinical and Radiological Findings
Brief Title: Irreparable Rotator Cuff Tears Treatment. Comparison of Two Methods: With and Without Biceps Tendon Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Lucas Hospital, Poland (Other)
Responsible Party: Principal Investigator, Hubert Laprus, Hubert Laprus, MD, Principal investigator. Department of Orthopaedic Surgery, Saint Lucas Hospital, Poland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLukasH
Record Dates: First submitted 2021-06-23; First posted 2021-08-12 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Massive Rotator Cuff Tears; Rotator Cuff Injuries; Shoulder Pain Chronic
Keywords: Massive rotator cuff; Partial repair; biceps augmentation; shoulder arthroscopy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: 2 different groups. Differences in type of surgery Comparison of two ways of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with biceps augmentation (Active Comparator): Complete repair of ISP if possible with partial SSP repair and biceps augmentation after its tenodesis
  Interventions: Procedure: Arthroscopic partial repair of rotator cuff with biceps augmentation
- Treatment without biceps augmentation (Active Comparator): Complete repair of ISP if possible with partial SSP repair and biceps tenotomy
  Interventions: Procedure: Arthroscopic partial repair of massive rotator cuff tear

INTERVENTIONS:
Procedure: Arthroscopic partial repair of massive rotator cuff tear — Surgery relies on arthroscopic reconstruction of the rotator cuff tendons. Because of irreparability of Supraspinatus tendon ( always) and infraspinatus tendon ( sometimes) surgeon performed partial repair to cover humeral head by the tendons
  Arms: Treatment without biceps augmentation
Procedure: Arthroscopic partial repair of rotator cuff with biceps augmentation — Surgery relies on arthroscopic reconstruction of the rotator cuff tendons. Because of irreparability of Supraspinatus tendon ( always) and infraspinatus tendon ( sometimes) surgeon performed partial repair to cover humeral head by the tendons and because of good quality of the long head of the biceps tendon, its uses as biological reinforcement of the reconstruction to achieve better clinical and radiological outcome
  Arms: Treatment with biceps augmentation

SUMMARY:
Management of massive rotator cuff tears (MRCT) is associated with high rates of failure. The long head of the biceps tendon augmentation (LHBTA) by reinforcement of the reconstruction and additional blood supply may improve healing and provide better outcome than partial repair only.

DETAILED DESCRIPTION:
Patients with irreparable supraspinatus muscle (SSP) tear, and complete infraspinatus muscle (ISP) tear are including in the prospective, comparative study. Excluding criteria consist of: problems or previous surgery of contralateral shoulder, subscapularis muscle tear larger than stage 2 by Lafosse classification, uncontrolled diabetes and previous surgery. First group consisting of patients treated by partial cuff repair with LHBTA. Second group is comparative group consisting of patients treated by only partial cuff repair without LHBTA. Group stratification depends on quality of the biceps tendon. In case of good tendon quality - its used for biological augmentation, if it's degenerated- tenotomy of the tendon and only partial repair is performing. Irreparability is defined as SSP ≥ 3 in Goutallier classification and stage 3 in Patte classification what is preoperatively assessed by MRI. Assessment tools consisting of range of motion (ROM), strength measurements in position adequate to assess reconstructing tendons and muscles force, Acromio-humeral index (AHI), Constant, SST, Hamada, and Sugaya scores. Goutallier classification for SSP and ISP and diameter of the teres minor muscle (TMn). Radiological and clinical assessment is performing one year after the surgery

ELIGIBILITY:
Inclusion Criteria:

Massive and irreparable rotator cuff tear:

* chronic supraspinatus tear with retraction grade 3 and muscle fatty infiltration ( measured in MRI ) > 3*
* Infraspinatus tear with retraction and fatty muscle degeneration

Exclusion Criteria:

* Previosus surgery
* Imposibility to performed MRI
* Diabetes
* no compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Comparison of improvement in shoulder range of motion | Through study completion, an average of 2.5 years
  Range of motion ( ROM) of every patient is measured preoperatively and postoperatively using goniometer and the result is presented in degrees. Comparision of two methods will be perform to assess better method for ROM improvement
Comparison of improvement in shoulder strength | Through study completion, an average of 2.5 years
  Strength will be measured by dynamometer in Kilograms [Kg] by main investigator in external rotation position, flexion, abduction and Jobe test position for every patient at the end of the study. Comparison of two methods will be perform to assess better method for shoulder strength improvement
Comparison of improvement in shoulder pain in VAS score | Through study completion, an average of 2.5 years
  Pain is assessed preoperatively and postoperatively using VAS score ( from 0 to 10, when 0 is no pain and 10 is the higher possible pain). Comparison of two methods will be perform to assess better method for shoulder pain reduce.
Comparison of shoulder function measured in Constant-Murley Score | Through study completion, an average of 2.5 years
  Function of the shoulder will be assess by Constant Murlay score which describes shoulder function in daily routines: In this score range is 0-100 when 100 is the best result.
Comparison of shoulder function measured in SST Score | Through study completion, an average of 2.5 years
  Function of the shoulder will be assess by SST score which describes shoulder function in daily routines: In this score range is 0-100% when 100% is the best result.

SECONDARY OUTCOMES:
Comparison of radiological outcome in Hamada score | Through study completion, an average of 2.5 years
  Radiological outcome will be assessed by Hamada score. This score measure shoulder cuff arthropathy ( stage 1-5 when 1 is the best result). For every patient this score will be calculated through study completion and comparison of two methods will be performed.
Comparison of radiological outcome in Sugaya score | Through study completion, an average of 2.5 years
  Radiological outcome will be assessed by Sugaya score. This score is used to measure quality of tendon reconstruction in MRI view. Range of points in this score is 1-5 when 1 is the best result. For every patient this score will be calculated through study completion and comparison of two methods will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Brzoska, Ph.D, MD, Study Chair — St Lukes's Hospital
Locations (1):
- Laprus, Bielsko-Biala, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No